CLINICAL TRIAL: NCT07055308
Title: Multisensory Patch to Measure Healthy and Abnormal Surgical Incision Healing
Acronym: SEASLUG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stichting IMEC-NL (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IM-NL-STUDY-2022-0028; CIV-23-06-043226 (Other: FAGG)
Record Dates: First submitted 2025-04-03; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Abdominal Surgery Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SeaPatch (Experimental): Daily measurement with multisensory patch from day 1 post-surgery maximally up to the day of discharge from hospital.
  Interventions: Device: SEAPatch

INTERVENTIONS:
Device: SEAPatch — Daily measurement with multisensory patch from day 1 post-surgery maximally up to the day of discharge from hospital.

SUMMARY:
Abdominal surgical incisions often lead to superficial surgical site infection (SSI). SSI is characterized by heat (calor), pain (dolor), redness (rubor), and swelling (tumor). The aim of this study is to measure calor, rubor and tumor with electronic sensors. Therefore, a multisensory patch is proposed which measures the tissue surrounding the incision once per day.

ELIGIBILITY:
Inclusion Criteria:

* The subject requires acute abdominal surgery due to perforation of the intestinal tractus (i.e., contamination upfront).
* The subject's incision is closed with either sutures or staples (by primary intention).
* The subject is 18 years or older.
* The subject can understand the patient information/ consent form and is capable of making his/her own decision.
* The subject is accompanied by an acquaintance who can give the second consent.

Exclusion Criteria:

* The subject has a known allergy to (silicon) adhesives.
* The subject states to be pregnant or planning to become pregnant.
* The subject receives medication that is contraindicated to excessive light exposure (e.g. Tetracylines, Doxycycline, Phenothiazines, Dacarbazine, Ketoprofen, Lomefloxacin). This criterion will be implemented in order to exclude the possibility of local skin irritation from prolonged irradiation by LED-light.
* The subject has an implantable device with a battery (i.e. pacemaker or other active implant).
* The subject has tattoos on the abdomen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-10-22 (Actual)

PRIMARY OUTCOMES:
Skin temperature around the surgical incision. | From day 1 post-operative up to 14 days post-operative
  Skin Temperature in degrees Celsius at multiple locations around the incision.
Bioimpedance around the incision. | From day 1 post-operative up to 14 days post-operative
  Bioimpedance in resistance and reactance at multiple locations around the incision.
PPG around the surgical incision. | From day 1 post-operative up to 14 days post-operative
  Reflective PPG in 3 different wavelengths around the surgical incision.

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuis Oost Limburg, Genk, Belgium